CLINICAL TRIAL: NCT03592238
Title: Sympathetic Nervous System Mediation of Acute Exercise Effects on Childhood Brain and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chuck Hillman, Professor, Northeastern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01HD094054-01 (NIH); R01HD094054 (NIH)
Record Dates: First submitted 2018-06-12; First posted 2018-07-19 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Exercise; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Psychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Intervention (Experimental): Participants will exercise on a motor-driven treadmill at a constant speed during the 23-min period.
  Interventions: Other: Aerobic Exercise Intervention
- Trier Social Stress Test for Children (Active Comparator): The Trier Social Stress Test for Children consists of a speech task in which children must finish a story and a mental arithmetic task, completed in front of a camera and two neutral observers.
  Interventions: Other: Trier Social Stress Test for Children
- Seated Rest (Placebo Comparator): Participants will sit in a comfortable chair, placed in the same room as the motor-driven treadmill, for a period of 25-min.
  Interventions: Other: Seated Rest

INTERVENTIONS:
Other: Aerobic Exercise Intervention — The protocol will include a 25-min bout of exercise at an intensity of 75% HRmax, such that participants will engage in a 1-min warm up and a 1-min cool down, with the majority of time (i.e., 23-min) spent exercising at 75% of HRmax.
  Arms: Aerobic Exercise Intervention
Other: Trier Social Stress Test for Children — Participants will be asked to imagine that they are in a new class with 20 other students, and that their teacher has asked them to stand in front of the class and introduce themselves. The mental arithmetic task will entail asking children to serially subtract the number 5 from a larger number as quickly as possible.
  Arms: Trier Social Stress Test for Children
Other: Seated Rest — Children will be asked to sit quietly or read a book of their choosing.
  Arms: Seated Rest

SUMMARY:
Today's children have become increasingly inactive and unfit, with >50% of children not meeting the recommended 60 min of moderate-to-vigorous physical activity. Previous research has suggested that acute aerobic exercise of moderate intensity was associated with improved cognition manifested by improved performance and increased P3 amplitude, a neuroelectric indicator that reflects the amount of attentional allocation, in tasks requiring cognitive control. While minimal evidence exists to support potential mechanisms underlying the transient effects of exercise on brain and cognition, research suggests that phasic changes in the locus coeruleus-norepinephrine (LC-NE) (as measured by salivary alpha amylase (sAA)) system are a potential mechanism for explaining the acute effect of exercise on brain and cognition. Accordingly, the aim of this study is to examine the mechanisms linking acute aerobic exercise to improved cognitive control as well as the underlying neuroelectrical activities in children, using electroencephalography (EEG) and event-related potentials (ERPs). We hope to gain a better understanding of the role of acute exercise and cognitive and brain health. The results from this study will help identify mechanisms linking acute exercise to enhanced cognitive performance in children.

Our hypothesis is that exercise-induced phasic increases in sympathetic nervous system activity will mediate the effect of a single bout of exercise on brain function, cognition, and standardized achievement test performance.

ELIGIBILITY:
Inclusion Criteria:

* Parental/guardian consent (non-consent of guardian).
* Participants must have had no prior diagnosis of cognitive or physical disability, including attention deficit hyperactivity disorder (severe asthma, epilepsy, chronic kidney disease, and dependence upon a wheelchair/walking aid).
* Participants must be free of any type of anti-psychotic, anti-depressant, anti-anxiety medication, as well as those medications used for attention deficit hyperactivity disorder (use of any anti-psychotic, anti-depressant, anti-anxiety, and attention deficit hyperactivity disorder medications).
* Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision).
* Participants must have not yet reached, or be in the earliest stages, of puberty, as measured by a modified test of the Tanner Staging System (onset of puberty as determined by Tanner).
* English speaking.

Exclusion Criteria:

* Participants with an intelligence quotient below 85 will be excluded.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Neuroelectric outcome | baseline
  P3 - ERP
Neuroelectric outcome | ~1 hr after arriving at lab, after completing the experimental condition
  P3 - ERP
inhibitory control | baseline
  accuracy
inhibitory control | baseline
  reaction time
working memory | baseline
  accuracy
working memory | baseline
  reaction time
inhibitory control | ~1 hr after arriving at lab, after completing the experimental condition
  accuracy
inhibitory control | ~1 hr after arriving at lab, after completing the experimental condition
  reaction time
working memory | ~1 hr after arriving at lab, after completing the experimental condition
  accuracy
working memory | ~1 hr after arriving at lab, after completing the experimental condition
  reaction time
Academic Achievement outcome | ~1.5 hrs after arriving at lab, after completing the experimental condition
  WRAT3 (Wide Range, Inc., Wilmington, DE) Reading Accuracy
Academic Achievement outcome | ~1.5 hrs after arriving at lab, after completing the experimental condition
  WRAT3 (Wide Range, Inc., Wilmington, DE) Spelling Accuracy
Academic Achievement outcome | ~1.5 hrs after arriving at lab, after completing the experimental condition
  WRAT3 (Wide Range, Inc., Wilmington, DE) Math Accuracy

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lloyd KM, Gabard-Durnam L, Beaudry K, De Lisio M, Raine LB, Bernard-Willis Y, Watrous JNH, Whitfield-Gabrieli S, Kramer AF, Hillman CH. Cross-sectional analysis reveals COVID-19 pandemic community lockdown was linked to dysregulated cortisol and salivary alpha amylase in children. Front Public Health. 2023 Dec 15;11:1210122. doi: 10.3389/fpubh.2023.1210122. eCollection 2023. PMID 38169630
- [Derived] Raine LB, Erickson KI, Grove G, Watrous JNH, McDonald K, Kang C, Jakicic JM, Forman DE, Kramer AF, Burns JM, Vidoni ED, McAuley E, Hillman CH. Cardiorespiratory fitness levels and body mass index of pre-adolescent children and older adults during the COVID-19 pandemic. Front Public Health. 2023 Jan 17;10:1052389. doi: 10.3389/fpubh.2022.1052389. eCollection 2022. PMID 36733279
- [Derived] Raine LB, McDonald K, Shigeta TT, Hsieh SS, Hunt J, Chiarlitti NA, Lim M, Gebhardt K, Collins N, De Lisio M, Mullen SP, Kramer AF, Hillman C. Sympathetic Nervous System and Exercise Affects Cognition in Youth (SNEACY): study protocol for a randomized crossover trial. Trials. 2021 Feb 18;22(1):154. doi: 10.1186/s13063-021-05096-w. PMID 33602325